CLINICAL TRIAL: NCT02621138
Title: The Influence of Muscle Contraction on the Cardiac Autonomic System at Rest and Activity
Brief Title: The Influence of Muscle Contraction on the Cardiac Autonomic System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 283-15
Record Dates: First submitted 2015-12-02; First posted 2015-12-03 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2015-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- cerebral palsy: Age 6-12 years Gross Motor Function Classification System I-II
- control: Age 6-12 years

SUMMARY:
Population:

16 children with cerebral palsy, GMFCS 1-3.16 children typically developed, matched for age.

All children aged 6-12 yrs who understand simple commands.

Tools:

1. Polar monitor to record heart rate, attached to chest, in use throughout testing
2. Dynamometer- for assessing muscle strength.
3. Weights

Method:

Each child will be tested once. Both tools will be demonstrated and tried out before actual testing.

With Polar watch attached:

1. 5 min sitting at rest,
2. knee muscle strength assessment with the dynamometer,
3. 15 minutes rest
4. Isometric and isotonic knee muscle contraction at 30% of childs' maximal strength as has assessed by the dynamometer. The child will asked to perform each for 3 minutes, with 5 minutes rest in-between All will be perform in both legs.

ELIGIBILITY:
Inclusion Criteria:

* GMFCS I-II
* Unilateral CP

Exclusion Criteria:

* Heart problems

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Heart rate | 40 minutes
Heart rate variability | 40 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Alyn Children's Rehabilitation Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided